CLINICAL TRIAL: NCT01818076
Title: Open Label Study to Assess Long-term Safety of Repeat Administration of Botulinum Toxin Type A for Moderate to Severe Crow's Feet Lines
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate study (not due to safety reasons)
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT001-CL023
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Skin Aging
MeSH Terms: interventions — Botulinum Toxins, Type A

ARMS (1):
- Dose A (Experimental): Dose A: Botulinum toxin type A
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botulinum toxin type A, Dose A applied to the lateral canthal area

SUMMARY:
This study will evaluate the long-term safety of botulinum toxin type A for the treatment of moderate to severe crow's feet lines after repeat application.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe crow's feet lines
* Female or male, 18 years of age and above and in good general health
* Women of childbearing potential must agree to use an effective method of birth control during the course of the study

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active skin disease or irritation at the treatment area
* Deep dermal scarring, or inability to smooth out the crow's feet lines to be treated by manually spreading the skin apart
* Treatment with botulinum toxin type A for crow's feet lines in the last 3 months
* Chemical peel during the 9 months prior to treatment
* Use of prescription retinoid products during the 3 months prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidences of treatment-emergent adverse events and serious treatment-emergent adverse events when the drug product is administered in repeated treatments | Up to 24 months
Incidences of treatment-emergent laboratory, skin erythema, cranial nerve, and ocular irritation abnormalities when the drug product is administered in repeated treatments | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee, United States